CLINICAL TRIAL: NCT04448418
Title: Observational Evaluation of the Impact of COVID-19 Outbreak on Transgender Subject's Health and on the Organization of Trans-population Health Care Services
Brief Title: The Impact of COVID-19 Outbreak on Trans-population's Health in Italy
Status: Completed | Type: Observational
Sponsor: Unita Complessa di Ostetricia e Ginecologia (Other)
Responsible Party: Principal Investigator, maria cristina meriggiola, Professor, Unita Complessa di Ostetricia e Ginecologia
Other Study IDs: TRANSCOVID-19
Record Dates: First submitted 2020-06-01; First posted 2020-06-25 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Transgender Persons; Coronavirus; Coronavirus Infection; COVID; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: web based survey — Assess specific health care needs for the transpopulation during the COVID-19 outbreack using a newly created questionnaire and some validated questionnaries (Impact of Event Scale-Revised, BECK Depression Inventory and the Self-rated Health SF-12)

SUMMARY:
During the COVID-19 outbreak, it was necessary to remodel the healthcare offer for all categories of subjects in order to minimize unnecessary movements of people while maintaining an adequate level of assistance. This is also true for transgender people, who are periodically requested to come into the clinic for hormonal therapy monitoring and continuation. In our center telemedicine programs dedicated to users have been activated for the remote management of hormone therapy.

We use a web-based survey to assess the impact of COVID-19 outbreak on trans-population health and to assess the specific needs of this population in this particular moment.

DETAILED DESCRIPTION:
Use of a dedicated web-based anonymous questionnaire to assess health needs of trans-population during COVID-19 outbreak and to assess specific risk factors for COVID-19 infection.

Evaluation of physical and psychological wellbeing of the trans-population during COIVD-19 outbreak in Italy using anonymous validated questionnaires (SF12, IES-R and BECK DEPRESSION INVENTORY)

ELIGIBILITY:
Inclusion Criteria:

* transgender subjects
* age > 18 years

Exclusion Criteria:

- none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: transgender population
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Assessment of the specific health need of the transpopulation during the COVID-19 pandemic in Italy | through study completion, an average of 6 months
  Evaluation of the specific health care needs of this population
Assessment of risk factors for COVID-19 infection in the traspopulation | through study completion, an average of 6 months
  Evaluation of socioeconomical and working condition of this population

SECONDARY OUTCOMES:
Evaluation of the satisfaction of this population with telemedicine for hormonal treatment monitoring | through study completion, an average of 6 months
  Use of a web based questionnaire to assess satisfaction with health care with a 0-10 scale (0=no satisfaction to 10=high satisfaction)
Evaluation of the psychological wellbeing of the trans-population during COVID-19 outbreak in Italy | through study completion, an average of 6 months
  Use of web based validated questionnaire: Impact of Event Scale-Revised (in Italian) to investigate perception of the COVID-19 event and subjects' mood. The scale is a self-report measure of current subjective distress in response to a specific traumatic event. Minimum score=0, maximum score=60, higher scores correspond to a worse outcome.
Evaluation of the psychological and physical wellbeing of the trans-population during COVID-19 outbreak in Italy | through study completion, an average of 6 months
  Use of web based validated questionnaire: Beck Depression Inventory to investigate mood. The 21 symptoms and attitudes contained in the questionnaire reflect the severity of the depression; the final score ranges from 0 to 63, with worse outcome with higher values.
Evaluation of the psychological and physical wellbeing of the trans-population during COVID-19 outbreak in Italy | through study completion, an average of 6 months
  Use of web based validated questionnaire: Short Form 2, to assess the impact of health on an individual's everyday life. The SF-12 is made of an eight-scale profile of scores as well as physical and mental health summary measures. Total scores range from 16 to 47 with worse outcomes for lower scores.

CONTACTS AND LOCATIONS:
Locations (1):
- 1Gynecology and Physiopathology of Human Reproduction, S. Orsola-Malpighi Hospital, Department of Medical and Surgical Sciences (DIMEC), University of Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No